CLINICAL TRIAL: NCT01930071
Title: PQ Bypass Guide Wire Delivery System for Femoropopliteal Bypass
Acronym: PQB4FP1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Endologix (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STP 114
Record Dates: First submitted 2013-08-20; First posted 2013-08-28 (Estimated); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PQ Bypass Guide Wire Delivery System (Experimental): PQ Bypass Guide Wire Delivery System to complete percutaneous Fem-pop bypass
  Interventions: Device: PQ Bypass Guide Wire Delivery System

INTERVENTIONS:
Device: PQ Bypass Guide Wire Delivery System — The PQ Bypass Guide Wire Delivery System is used to bypass lesions in the peripheral vasculature percutaneously. A guidewire is placed from the artery proximal to the lesion to the artery distal to the lesion using the vein as a conduit with the Guidewire Delivery System. Once in place, commercially available stent grafts will be placed to complete the bypass.

SUMMARY:
To assess the safety of performing a percutaneous fem-pop bypass using the PQ Bypass Guidewire Delivery System and commercially available stent grafts.

DETAILED DESCRIPTION:
Multi-center, single-arm first-in-man study utilizing the PQ Bypass Guide Wire Delivery System to access, deliver guidewires and implant stent grafts for a percutaneous femoropopliteal (fem-pop) bypass.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide informed consent
* Age 18 or older
* Rutherford Classification of 3-5
* Lesions ≥10cm in length considered to be:

  * Chronic total occlusion (100% stenosis)
  * Diffuse stenosis (>50% stenosis) with moderate to heavy calcification
  * In-stent restenosis (>50% stenosis)
* Proximal and distal target vessels are 4.8 - 7.5 mm in diameter
* Orifice and proximal 1cm of SFA is patent
* Patent popliteal artery 3cm proximal to tibial plateau
* At least 1 patent tibial artery to the foot
* Patent femoral vein

Exclusion Criteria:

* History of deep vein thrombosis
* Has a known sensitivity or allergy to contrast materials that cannot be adequately pre-treated
* Has a known sensitivity or allergy to aspirin, heparin or anti-platelet medications
* Documented in-sensitivity to anti-platelet medication
* Has a known or previous coagulopathy
* Pregnant or lactating
* Untreated flow-limiting aortoiliac occlusive disease
* Has renal failure (GFR < 30mL/min)
* Major distal amputation (above the transmetatarsal) in the study or non-study limb
* Patient has had a procedure on the target limb within 30 days
* Previous bypass surgery on the target limb
* Bypass length required is greater than 35cm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2013-11; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Primary Patency | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Holden, MD, Principal Investigator — Auckland City Hospital
Locations (1):
- Auckland City Hospital, Auckland, New Zealand